CLINICAL TRIAL: NCT04762355
Title: A Phase 1, Double-Masked, Vehicle-Controlled Study to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Palovarotene Ophthalmic Solution in Healthy Adult Subjects
Brief Title: Study to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Palovarotene Ophthalmic Solution in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVO-3A-101
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Palovarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): Subjects were randomized in a 3:1 ratio to receive one dose regimen of either active treatment or placebo (vehicle). Advancement of the study from the once daily (QD) dosing regimen to the twice daily (BID) dosing regimen, and dose escalation to the next dose regimen
  Interventions: Drug: Palovarotene; Drug: Vehicle
- Dose 2 (Experimental): Subjects were randomized in a 3:1 ratio to receive one dose regimen of either active treatment or placebo (vehicle). Advancement of the study from the once daily (QD) dosing regimen to the twice daily (BID) dosing regimen, and dose escalation to the next dose regimen
  Interventions: Drug: Palovarotene; Drug: Vehicle
- Dose 3 (Experimental): Subjects were randomized in a 3:1 ratio to receive one dose regimen of either active treatment or placebo (vehicle). Advancement of the study from the once daily (QD) dosing regimen to the twice daily (BID) dosing regimen, and dose escalation to the next dose regimen
  Interventions: Drug: Palovarotene; Drug: Vehicle

INTERVENTIONS:
Drug: Palovarotene — ophthalmic solution in different concentrations: Dose 1, Dose 2 and Dose 3
Drug: Vehicle — Placebo-to-match palovarotene ophthalmic solution vials

SUMMARY:
Dry eye disease (DED) is a keratoconjunctive disorder that "is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. The goal of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of multiple ascending doses of palovarotene ophthalmic solution in healthy adult subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, male or female, 18 to 55 years of age, inclusive, at screening.
* Continuous non-smoker who had not used nicotine containing products for at least 3 months prior to the first dosing and throughout the study, based on subject self-reporting.
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m2 at screening.
* Medically healthy as deemed by the Investigator or delegate and determined by medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory results obtained within 28 days before the start of the study.
* Tolerate topical administration to the eye.
* Best corrected visual acuity is equal or better than 70 Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in both eyes.

Key Exclusion Criteria:

* Mentally or legally incapacitated or had significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical (systemic or ophthalmic) or psychiatric condition or disease in the opinion of the Investigator or delegate.
* History of any illness that, in the opinion of the Investigator or delegate, might have confounded the results of the study or posed an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 18 months prior to the first dosing.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug, systemic retinoids such as isotretinoin or related compounds (e.g., topical tretinoins, vitamin A), fluorescein, or parabens or to the inactive ingredients in the study formulation.
* History of any ocular surgery or laser within the past 6 months prior to screening.
* History of herpes simplex keratitis.
* History or presence of:

  1. Any chronic eye disease other than refractive error, incipient cataract, strabismic amblyopia, or anisometropic amblyopia.
  2. Acute eye disease (such as infection, corneal abrasion, or allergy) within the past 6 months from screening.
* Any currently active ocular condition that required use of topical eye drops.
* Had an intraocular pressure >21 mmHg.
* If ophthalmological examination at screening or Day 1 predose revealed abnormalities of the cornea, evidence of ocular infection, inflammation (dry eyes, blepharitis, allergic conjunctivitis, iritis, and uveitis), advanced or moderately injected pterygium, keratitis, narrow anterior chamber angles, clinically significant Meibomian gland dysfunction, or any finding in either the anterior segment or posterior segment of the eye, that could have compromised the study as per Investigator or delegate discretion.
* Any macular integrity issues or optic nerve head (ONH) cupping/abnormality on retinal exam.
* Occurrence of active seasonal allergies including ocular allergies (e.g., annual hay fever).
* Needed to wear contact lenses during the study.
* Positive results at screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus.
* Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study, unless permitted by the Investigator or delegate.
* Any drugs known to be significant inhibitors and inducers of CYP3A4 enzymes, including St. John's Wort, for 30 days prior to the first dosing and throughout the study.
* Ocular medication of any kind (including artificial tears), antihistamines, anticholinergics, and/or oral/nasal steroids for 30 days prior to the first dosing and throughout the study.
* Isotretinoin or other systemic retinoids beginning 30 days or 5 half-lives, whichever was longer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent ocular adverse events (TEAEs) | from baseline until the end of study (up to 25 days)
Change in ocular safety measurements as determined by Best-Corrected Visual Acuity (BCVA) | from baseline until the end of study (up to 25 days)
Change in Corneal Fluorescein Staining | from baseline until the end of study (up to 25 days)
Change in intraocular pressure | from baseline until the end of study (up to 25 days)

SECONDARY OUTCOMES:
Plasma concentration (predose) observed at the end of a dosing interval (Ctrough) | Day 5 and Day 6 (prior to the morning), Day 7 ((prior to the morning), Day 8, Day 9, Day 10
Area under the concentration-time curve during a dosing interval (AUCtau) | Day 7 and Day 10
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) | Day 10
Maximum observed concentration at steady state (Cmax,ss) | Day 7 and Day 10
Average concentration at steady state (Cavg) | Day 7 and Day 10
Apparent total plasma clearance after topical administration (CL/F) | Day 7 and Day 10
Time to reach Cmax at steady state (Tmax) | Day 7 and Day 10
Apparent first-order terminal elimination half-life (t½) | Day 7 and Day 10
Apparent first-order terminal elimination rate (k el) | Day 7 and Day 10
Apparent volume of distribution (Vss/F) | Day 7 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Algorithme Pharma facility, Québec, Canada